CLINICAL TRIAL: NCT03118973
Title: Evaluation of Efficacy and Safety of Goff Transpancreatic Septotomy vs. Double Wire Technique for Achieving Biliary Access in Technically Challenging ERCPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Subhas Banerjee (Other)
Responsible Party: Sponsor-Investigator, Subhas Banerjee, Associate Professor of Medicine, Division of Gastroenterology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38574
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Biliary Obstruction; Biliary Stones
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Intervention Model Description: Patients with challenging biliary cannulation randomized to either Goff trans-pancreatic septotomy or double wire technique to facilitate biliary cannulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goff (Experimental): For patients in whom biliary cannulation is difficult to achieve, Goff trans-pancreatic septotomy will be performed to facilitate biliary cannulation.
  Interventions: Procedure: Goff trans-pancreatic septotomy vs. Double wire technique
- Double wire (Experimental): For patients in whom biliary cannulation is difficult to achieve, double wire technique will be used to facilitate biliary cannulation.
  Interventions: Procedure: Goff trans-pancreatic septotomy vs. Double wire technique

INTERVENTIONS:
Procedure: Goff trans-pancreatic septotomy vs. Double wire technique — Goff trans-pancreatic septotomy vs. Double wire technique for achieving biliary access when biliary cannulation is challenging.

SUMMARY:
Randomized, prospective study evaluating efficacy and safety of Goff transpancreatic septotomy vs. double wire technique for achieving biliary access in patients who fail initial cannulation at ERCP.

DETAILED DESCRIPTION:
Selective placement of a guidewire into the bile duct (biliary cannulation) during endoscopic retrograde cholangiopancreatography (ERCP) is necessary for performing therapeutic biliary procedures. The success rate for biliary cannulation by experienced endoscopists during ERCP is approximately 85% with standard cannulation techniques. Inadvertent placement of the guidewire into the pancreatic duct rather than the bile duct often occurs when attempting selective biliary cannulation in technically challenging cases. When this occurs repeatedly, other approaches may be used to facilitate selective biliary cannulation, but there are few prospective studies evaluating the efficacy and safety of these approaches. Here the investigators evaluate two approaches for technically challenging biliary cannulation: one involving maintenance of a wire in the pancreatic duct, followed by repeat attempt at biliary cannulation (double wire technique) and one involving a small incision in the septum adjacent to the pancreas followed by repeat attempt at biliary cannulation (transpancreatic septotomy). This study is a prospective randomized trial comparing the rate of cannulation success, procedure duration and complications following these two approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Patient has a clinical indication for ERCP
3. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Age <18
2. Potentially vulnerable subjects including, homeless people, pregnant females, employees and students.
3. Complex post-surgical anatomy e.g. Billroth type II anatomy, Roux-en-Y-gastrojejunostomy
4. Prior sphincterotomy or balloon dilation of ampulla
5. Thrombocytopenia, coagulopathy, or indication for ongoing anti-coagulation therapy
6. Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Successful biliary cannulation assessed by fluoroscopic confirmation of biliary cannulation | Day of procedure
  Successful biliary cannulation

SECONDARY OUTCOMES:
Adverse event rates assessed by 6-month follow-up of clinical and laboratory studies | 6 months
  Rates of adverse events associated with the ERCP procedure following intervention to facilitate biliary cannulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No